CLINICAL TRIAL: NCT05914506
Title: Hyperpolarized 129-Xenon MRI in Fibrosing Interstitial Lung Disease
Status: Active, not recruiting | Type: Observational
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Xe-F-ILD-001; 2022-502512-36-00 (Other: European Medicines Agency (EU CT)); U1111-1284-7436 (Registry Identifier: Universal Trial Number (WHO))
Record Dates: First submitted 2022-11-10; First posted 2023-06-22 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Progressive Fibrosing Interstitial Lung Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: Hyperpolarized xenon-129 MRI — Participants will be asked to inhale the xenon-129 contrast agent according to procedure for gas administration. The success criterion of the drug is a obtained Xe MRI lung image with reasonable signal level

SUMMARY:
This project aims to investigate the potential of non-invasive imaging to identify and monitor the earliest signs and physiological effects of pulmonary fibrosis and resulting cardiac dysfunction in patients with fibrosing interstitial lung disease. Second, to evaluate baseline risk factors the progression and therapeutic responses to anti-fibrotic drugs.

DETAILED DESCRIPTION:
Fibrosing interstitial lung diseases (F-ILD) represent a heterogeneous disease category involving several disease entities with different clinical, radiological, and histological characteristics. The common denominator for F-ILD patients is similarities regarding development of scarring of the lungs. Idiopathic pulmonary fibrosis (IPF) is the prototype, and all patients will eventually suffer from irreversible progression. In other type of F-ILD, a proportion of patients will also develop symptom worsening, treatment resistance towards immunomodulatory therapy, a decline in lung physiological parameters, worsening of radiologic findings and irreversible self-sustaining progression of pulmonary fibrosis i.e., a phenotype of progressive pulmonary fibrosis (PPF), defined by worsening of symptoms, lung physiology and radiology within 12 months Chest High Resolution Computed Tomography (HRCT) is considered the golden standard to diagnose and quantify the type and extent of pulmonary fibrosis. Extent of fibrosis and specific features like traction bronchiectasis and honeycombing seem in some disease to be associated with a worse outcome. However, findings do not always correspond to disease severity or disease course, and at later stages, HRCT is limited in proving the progression of the disease. Identifying progression is currently based on a decrease in forced vital capacity (FVC), diffusing capacity for carbon monoxide (DLCO), worsening of symptoms or progression of radiologic features (Table 1). Identification of radiologic biomarkers for progression will allow to better support treatment decisions and inform patients. Patients with F-ILD often suffer from a high burden of comorbidities, including ischemic heart disease, congestive heart failure, and pulmonary hypertension. It is currently unknown if these is solely associated to common risk factors like smoking and age, or could be due to fibrosis developing in the myocardium. Furthermore, it is not well described if the development of a restrictive lung physiology plays a role and affects cardiac physiology.

This study proposes that MR (magnetic resonance) Imaging with hyperpolarized 129Xenon will be able to detect subtle, regional dysfunction of the gas exchange of the lungs in patients with F-ILDs at a higher level of sensitivity than currently applied techniques. Utilizing the improved sensitivity of the hyperpolarized xenon MRI the study aims to improve the diagnostic distinction between the different subtypes of F-ILDs and additionally point-out MR biomarkers to be assess F-ILD severity, progression, and potential treatment response. Simultaneously with the hyperpolarized 129Xe scans, imaging of myocardial strain and ejection fraction is performed. In addition, a Gadolinium Based Contrast Agent (GBCA) is administered to evaluate the degree of myocardial fibrous tissue and lung perfusion. Thus, the impact of thoracic restrictive physiology on the heart can be detected and quantified.

ELIGIBILITY:
Inclusion Criteria:

* Informed signed consent
* Age 18-90
* Pre-menopausal women must be confirmed non-pregnant by an onsite test.
* Patients diagnosed with IPF or fibrotic ILD who fulfills PPF criteria, and are prescribed antifibrotic treatment.
* Cognitively able to understand and participate in the study

Exclusion Criteria:

* Contraindications for MRI:

  * Pacemaker, neurostimulator or cochlear implant
  * Metal foreign bodies such as fragments and irremovable piercings
  * Unsafe medical implants (safety of heart valves, hips and the like must be confirmed)
  * Intrathoracic clips or coils
  * Cardiac pacemakers
  * Claustrophobia
  * Largest circumference including arms > 160 cm
* Contraindications to gadolinium contrast

  * eGFR < 30 mL/min/1.73m2
  * Previous adverse reactions to gadolinium
* Overlapping emphysemic disease where the emphysema-component outweighs the fibrosis
* Unable to perform breath-hold of minimum 20 seconds.
* Allergy to Xenon
* Breast feeding
* Evidence of ongoing respiratory infections at time of MR examinations

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have recently recieved a diagnosis of progressive fibrosing interstial lung disease and are expected to recieve antifibrotic therapy
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-10-05 (Actual); Primary Completion 2028-05-01 (Estimated); Study Completion 2028-05-01 (Estimated)

PRIMARY OUTCOMES:
Xenon gas transfer | 12 months
  Gas transfer across the lung barrier measured using dissolved phase Xe-129 gas MRI spectroscopy.
  From this measure we expect to see an increase in the tissue signal and a decrease in the blood signal as a measure of IPF disease activity.
  We expect the change in ratio to be more than 10% when comparing baseline results to follow-up at subject level.
  Results will be compared to clinical outcome measures of progression (outcome 2)
Individual clinical progression in the study period (progressors and non-progressors) | 12 months
  Current accepted criteria for progression of fibrosing interstitial lung diseases (at least 2 of 3):
  1. Worsening of clinical symptoms (estimated by qualified physician. Additionally this will be quantified by patient related outcome measures, (K-BILD, SOBQ and L-PF)
  2. Decline in pulmonary function test parameters (decrease of FVC >= 5% and/or DLCO >= 10%)
  3. Radiological evidence of disease progression:
     1. Increased extent or severity of traction bronchiectasis and bronchiolectasis
     2. New ground-glass opacity with traction bronchiectasis
     3. New fine reticulation
     4. Increased extent or increased coarseness of reticular abnormality
     5. New or increased honeycombing
     6. Increased lobar volume loss.

SECONDARY OUTCOMES:
Pulmonary perfusion | 12 months
  Regionally decreased pulmonary perfusion in ml/g/min measured by gadolinium enhanced MRI
Myocardial strain | 12 months
  Evidence of myocardial strain measured by relative myocardial deformation through the cardiac cycle in percentage with CINE MRI
Fibrous tissue formation | 12 months
  Formation of fibrotic tissue measured with late-contrast enhancement and evaluated as MRI signal intensity changes before and after intravenous gadolinium injection.
Xenon ventilation distribution | 12 months
  Ventilation defect is measured by xenon gas distribution in the lungs. Ventilation defect percentage is quantified by xenon MRI signal divided by whole lung volume.
Xenon gas diffusion | 12 months
  The diffusion of xenon gas in the alveoli. Gas diffusion is measured with diffusion-weighted xenon MRI as gas-molecule speed (cm/s)

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth Bendstrup, Professor, Principal Investigator — Aarhus University Hospital
Locations (1):
- Aarhus University, Department of Clinical Medicine, MR Research Centre, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No